CLINICAL TRIAL: NCT03116269
Title: The Effect of Cilostazol Compared to Aspirin on Endothelial Function Measured by Flow Mediated Dilatation in Acute Cerebral Ischemia Patients
Brief Title: The Effect of Cilostazol Compared to Aspirin on Endothelial Function in Acute Cerebral Ischemia Patients
Acronym: PASS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Man Hong, Associate proffessor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AJIRB MED CT4 10-239
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Ischemic Stroke; Endothelial Dysfunction
MeSH Terms: conditions — Ischemic Stroke | interventions — Cilostazol; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cilostazol group (Experimental): aspirin placebo daily and 100 mg cilostazol twice daily
  Interventions: Drug: Cilostazol 100mg
- aspirin group (Active Comparator): 100 mg aspirin daily and cilostazol placebo twice daily
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Cilostazol 100mg
  Arms: cilostazol group
Drug: Aspirin
  Arms: aspirin group

SUMMARY:
Patients presenting with acute cerebral ischemic events are randomly assigned into aspirin (n=40) or cilostazol (n=40) group in a double-blinded manner. FMD is measured as a primary outcome at baseline (T0) and 90 days (T1). Serious and non-serious adverse events were described.

DETAILED DESCRIPTION:
This investigator-initiated, randomized, double-blind trial is prospectively conducted with two-arm parallel treatment groups and a single dose scheme: 100 mg aspirin daily and cilostazol placebo twice daily versus aspirin placebo daily and 100 mg cilostazol twice daily.

A total of 80 eligible patients is planned to be recruited.

All included patients undergo diagnostic studies including routine blood tests and cardiologic work-ups. The primary outcome is differences in endothelial function in the two groups measured by means of FMD on admission and at 3 months. According to previous studies, the adverse effects in two groups are investigated.

ELIGIBILITY:
Inclusion Criteria:

1. acute ischemic stroke confirmed by diffusion weighted imaging
2. transient ischemic attack (TIA) within 7 days

Exclusion Criteria:

1. there is intracranial hemorrhage on imaging study
2. patients is previously taking antiplatelets, vitamin K antagonists, factor Xa antagonists, or chronic treatment with systemic steroidal and non-steroidal anti-inflammatory drugs
3. patients who received fibrinolytics within the previous 48 hours
4. cognitive impairment interfering with the possibility of obtaining informed consent
5. pregnancy
6. participation in another pharmacological study
7. peptic ulcer disease or hematological abnormality
8. initial modified Barthel index <30 points
9. liver function tests exceeding a 2-fold upper range value.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2014-10-31 (Actual)

PRIMARY OUTCOMES:
flow mediated dilation | 3 month change
  flow mediated dilation of the brachial artery in response to hyperemia

CONTACTS AND LOCATIONS:
Overall Officials: Ji Man Hong, Principal Investigator — 82 31 219 5174
Locations (1):
- Ajou University Medical Center, Suwon, Gyunggido, South Korea

REFERENCES:
- [Derived] Lee SJ, Lee JS, Choi MH, Lee SE, Shin DH, Hong JM. Cilostazol improves endothelial function in acute cerebral ischemia patients: a double-blind placebo controlled trial with flow-mediated dilation technique. BMC Neurol. 2017 Aug 29;17(1):169. doi: 10.1186/s12883-017-0950-y. PMID 28851320